CLINICAL TRIAL: NCT05786456
Title: Novel e-Health Intervention for Fear of Progression in Women With Gynecologic Cancer: A Pilot Study
Brief Title: e-Health Intervention (Day-by-Day) for the Management of Fear of Progression in Women With Stage III or IV Gynecologic Cancer: A Pilot Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 22683; NCI-2023-00309 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 22683 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2023-03-10; First posted 2023-03-27 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Malignant Female Reproductive System Neoplasm; Stage III Cervical Cancer AJCC v8; Stage III Ovarian Cancer AJCC v8; Stage III Uterine Corpus Cancer AJCC v8; Stage III Vaginal Cancer AJCC v8; Stage III Vulvar Cancer AJCC v8; Stage IV Cervical Cancer AJCC v8; Stage IV Ovarian Cancer AJCC v8; Stage IV Uterine Corpus Cancer AJCC v8; Stage IV Vaginal Cancer AJCC v8; Stage IV Vulvar Cancer AJCC v8
MeSH Terms: conditions — Uterine Cervical Neoplasms; Ovarian Neoplasms; Vaginal Neoplasms; Vulvar Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive Care (DBD) (Experimental): Patients receive DBD intervention consisting of group and web-based self-study sessions and check-in calls on study. Patients also watch videos and receive handouts to reinforce the group sessions.
  Interventions: Procedure: Discussion; Other: Informational Intervention; Other: Media Intervention; Other: Questionnaire Administration; Behavioral: Telephone-Based Intervention

INTERVENTIONS:
Procedure: Discussion — Participate in group and web-based self-study sessions
  Other Names: Discuss
Other: Informational Intervention — Receive handouts
Other: Media Intervention — View videos
Other: Questionnaire Administration — Ancillary studies
Behavioral: Telephone-Based Intervention — Participate in check-in calls

SUMMARY:
This clinical trial studies how well an electronic (e)-health intervention (day-by-day) woks in managing fears or worries about cancer growing, spreading, or getting worse (progression) in patients with stage III or IV gynecologic cancer. Fear and worries about cancer progression or recurrence (coming back) are common concerns. This may contribute to concerns related to illness, worries, and uncertainty about the future. Day by Day is adapted from a program called "Conquer Fear" which was shown to benefit patients with early-stage cancer. Day-by-day intervention may help refocus patient thoughts and help patients learn skills to manage anxiety and fears.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Will adapt the intervention into a hybrid format including two group and three web based self-study sessions. (Phase 1) II. To determine the feasibility and acceptability of a new hybrid e-health intervention to manage fear of progression (FOP) in patients with stage III or IV gynecologic (GYN) cancer. (Phase 2)

SECONDARY OBJECTIVE:

I. To explore the preliminary efficacy of day-by-day (DBD) on reducing FOP (primary outcome) and improving secondary outcomes of distress, anxiety, depression, metacognitions, and mindfulness. (Exploratory)

OUTLINE:

PHASE I (DEVELOPMENT): Patients complete surveys and participate in focus groups.

PHASE II (DBD): Patients receive DBD intervention consisting of group and web-based self-study sessions and check-in calls on study. Patients also watch videos and receive handouts to reinforce the group sessions.

ELIGIBILITY:
Inclusion Criteria:

* Women with stage III or IV GYN cancer (ovarian, endometrial, cervical, vulvar/vaginal);at least 3 months from initial diagnosis
* Age: >= 18 years
* Score >= 34 on the Fear of Progression Short-Form, indicating dysfunctional levels
* Ability to read and understand English
* Patients in remission or with progressive disease are eligible

Exclusion Criteria:

* Enrolled in hospice
* Severe depression as assessed by Patient Health Questionnaire (PHQ-9)
* Non-English speaking
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2024-07-19 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Feasibility of recruitment (enrollment rate) | Up to 6 weeks
  Defined by attendance, attrition, and skills practice adherence. Website acceptability is based on the System Usability Scale, log-in activity, activity completion rate, and most frequently visited site content.

SECONDARY OUTCOMES:
Fear of progression (FOP) | Up to 12 weeks
  FOP will be assessed using FOP Questionnaire-Short Form (SF) at baseline (T1), weeks (T2), and 12 weeks (T3). FOP-Q-SF consists of 12 items scored on a 5-point Likert scale (1=never to 5=very often); scores range from 12-60 with higher levels indicating greater FOP. Researchers have used a cut-off of 34 and above to indicate dysfunctional FOP.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Reb, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States